CLINICAL TRIAL: NCT05793580
Title: Long Term Results With the Vibrant Soundbridge in Patients With Mixed Hearing Loss: a Prospective Multicenter Longitudinal Study Over 60-months
Brief Title: Long Term Results With the Vibrant Soundbridge in Patients With Mixed Hearing Loss: a 60-month Longitudinal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VSB_longterm_Rennes_study
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Mixed Hearing Loss
Keywords: Active middle ear implant; Vibrant Soundbridge
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Intervention Model Description: Prospective longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VSB arm (Other): longitudinal follow-up of VSB users preoperatively and at 1, 3, 6, 12 and 60 months post-implantation.
  Interventions: Device: Vibrant Soundbridge active middle ear implant

INTERVENTIONS:
Device: Vibrant Soundbridge active middle ear implant — active middle ear implant

SUMMARY:
Vibrant Soundbridge (VSB, MED-EL, Innsbruck) Active middle ear implants (AMEI) can benefit patients who are unable to use conventional hearing aids (HA) due to medical reasons, discomfort or unsuccessful rehabilitation. Long-term prospective longitudinal studies are lacking on the VSB notably for conductive and mixed hearing loss. The main aim of the present study was to prospectively assess aided hearing benefits in a 60-month, long-term study including conductive and mixed hearing loss adults implanted with the VSB. The secondary objective was to compare the hearing results according to the Floating Mass Transducer (FMT) site (Round/oval window (RW/OW) vs incus/stapes) and the type of pathology responsible for the hearing loss (Inflammatory vs non-inflammatory disease, ID vs NID).

DETAILED DESCRIPTION:
Introduction:

Active middle ear implants (AMEI) can benefit patients who are unable to use conventional hearing aids (HA) due to medical reasons, discomfort or unsuccessful rehabilitation.

AMEIs provide more hearing gain and consistency compared to middle ear surgery plus conventional hearing aids. Coletti et al. (2013) reported on long-term outcomes of patients implanted at the round window (RW) with the VSB. Brkic et al. (2019) presented a large number of subjects (n = 23) with a 20-year follow-up. The limitations of these studies were their retrospective design.

The best location for the surgeon to place the VSB's floating mass transducer (FMT) depends on various factors. A meta-analysis showed the hearing results at different FMT sites to be similar. None of these studies compared a FMT placed to a FMT clipped.

The impact of the etiology of deafness on a patient's outcome with an AMEI has been poorly studied. Only one study has shown that the difference between inflammatory disease (ID) and non-inflammatory disease (NID) groups was not significant.

The main objective:

Prospectively assess aided hearing benefits in a 60-month, long-term study including conductive and mixed hearing loss adults implanted with the VSB.

Measures are tonal audiometry, pure-tone average (PTA), vocal audiometry in quiet, 50% speech recognition threshold (SRT) in quiet, word recognition in quiet (WRS) at 65 dB sound pressure level (SPL), word recognition in noise (WRSN ; speech at 65 dB SPL and 0°, white noise at 55 dB SPL and 180°. signal-to-noise ratio = 10 dB).

The secondary objectives:

Comparison of the hearing results according to the FMT site (RW/OW to incus/stapes)

Comparison of the hearing results according the type of pathology responsible for the hearing loss (ID to NID).

Plan of the study:

It is a multicentric, prospective, longitudinal study with 6 tertiary references centres with a follow up over a period of 60 months.

Measures will be done on the patient preoperatively and 1, 3, 6, 12 and 60 months post-implantation.

Preoperative measures will be done also with hearing aid (HA) and bone-anchored hearing aid on a headband (HBAHA).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* with mixed hearing loss on at least one side
* with a maximum bone conduction (BC) threshold of 45 dB hearing level (HL) at 500 Hz, 50 dB HL at 1000 Hz, 55 dB HL at 1500 Hz, and 60 dB HL at 2000 Hz.
* with a 20 dB minimum air-bone gap (defined as the difference between bone- and air conduction thresholds).
* with stable BC thresholds over the previous 24 months, and no sufficient benefit with the HA.

Exclusion Criteria:

* fluctuating hearing loss,
* cutaneous disease
* subjects who need an MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Tonal audiometry | preoperatively
  Pure-tone audiograms
Tonal audiometry | at 1 month post-implantation
  Pure-tone audiograms
Tonal audiometry | at 3 months post-implantation
  Pure-tone audiograms
Tonal audiometry | at 6 months post-implantation
  Pure-tone audiograms
Tonal audiometry | at 12 months post-implantation
  Pure-tone audiograms
Tonal audiometry | at 60 months post-implantation
  Pure-tone audiograms

SECONDARY OUTCOMES:
Word recognition in quiet | preoperatively
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in quiet | at 1 month post-implantation
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in quiet | at 3 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in quiet | at 6 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in quiet | at 12 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in quiet | at 60 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists).
Word recognition in noise | preoperatively
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Word recognition in noise | at 1 month post-implantation
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Word recognition in noise | at 3 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Word recognition in noise | at 6 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Word recognition in noise | at 12 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Word recognition in noise | at 60 months post-implantation
  Speech recognition test of disyllabic words (Fournier lists) in noise. Noise = white noise at 55 dB SPL presented at 180°. Speech at 65 dB SPL presented at 0°.
Speech reception threshold | preoperatively
  Speech reception threshold to have 50% of intelligibility on disyllabic words.
Speech reception threshold | at 1 month post-implantation
  Speech reception threshold to have 50% of intelligibility on disyllabic words.
Speech reception threshold | at 3 months post-implantation
  Speech reception threshold to have 50% of intelligibility on disyllabic words.
Speech reception threshold | at 6 months post-implantation
  Speech reception threshold to have 50% of intelligibility on disyllabic words.
Speech reception threshold | at 12 months post-implantation
  Speech reception threshold to have 50% of intelligibility on disyllabic words.
Speech reception threshold | at 60 months post-implantation
  Speech reception threshold to have 50% of intelligibility on disyllabic words.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Godey, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No